CLINICAL TRIAL: NCT06297018
Title: The Effect of Bioenergy Application
Brief Title: Bioenergy, Depression, Anxiety and Stress After Liver Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collect completed
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, SEMRA BÜLBÜLOĞLU, Clinical Associate Professor, Istanbul Aydın University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: February 18, 2024
Record Dates: First submitted 2024-02-18; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue
Keywords: Biyoenergy; anxiety; stress; liver transplant recipients
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Interventional Crossover Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (No Intervention): No intervention: This group includes liver transplant recipients and no intervention is applied to this group. Depression, anxiety and stress levels are measured in the pre-test. No intervention is implemented. As a post-test, depression, anxiety and stress levels are measured again.
- 2 (Experimental): Bioenergy group: This group includes liver transplant recipients and recipients who underwent intervention. Depression, anxiety and stress levels are measured in the pre-test. Bioenergy is then applied. As a post-test, depression, anxiety and stress levels are measured again.
  Interventions: Behavioral: Bioenergy application

INTERVENTIONS:
Behavioral: Bioenergy application — Bioenergy application: This group includes liver transplant recipients and recipients who underwent intervention. Depression, anxiety and stress levels are measured in the pre-test. Bioenergy is then applied. As a post-test, depression, anxiety and stress levels are measured again.
  Other Names: Bio fields
  Arms: 2

SUMMARY:
In this study, the investigators aimed to examine the effect of bioenergy application on depression, anxiety and stress after liver transplantation.

DETAILED DESCRIPTION:
Simple random sampling method was used to assign liver recipients to experimental and control groups. Discharged liver transplant patients will be investigated for anxiety, stress and depression.

ELIGIBILITY:
Inclusion Criteria:

(i) liver transplant recipient (ii) must be able to use immunosuppressive agents (iii) 18 years or older Liver transplant recipients

Exclusion Criteria:

having psychiatric problems having language and communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Anxiety, stress, depression: Measurement will be made with the Depression Anxiety Stress 21 Scale (DASS-21: Score range 21-63) | total of six month
  It will be measure Therapy on Liver Transplant Recipients'

CONTACTS AND LOCATIONS:
Locations (1):
- Semra Bulbuloglu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No